CLINICAL TRIAL: NCT04464382
Title: A Randomized Double-blind Clinical Trial to Evaluate the Safety and Efficacy of a Outpatient Appendectomy (PENDI_CSI)
Brief Title: Evaluating the Safety and Efficacy of a Outpatient Appendectomy
Acronym: PENDI_CSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PENDI_CSI
Record Dates: First submitted 2020-02-11; First posted 2020-07-09 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-07

CONDITIONS: Appendicitis Acute; Appendectomy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient appendectomy (Experimental): Patients with acute uncomplicated appendicitis that require emergency appendectomy. The intervention will be the classic.Once the appendectomy is performed, all the selection criteria will be reassessed and the definitive inclusion of the patients will be performed.
  Patients after surgery will go to the anesthetic recovery room without requiring hospital admission. The degree of satisfaction of the quality of the service and the care that must be completed before discharge and after surgery will be recorded.
  1 phone review call will be made per month +/- 30 days in order to assess the safety and satisfaction of the procedure.
  Interventions: Procedure: Outpatient (OA)
- Hospitalization appendectomy (Active Comparator): Patients with acute uncomplicated appendicitis that require emergency appendectomy. The intervention will be the classic.Once the appendectomy is performed, all the selection criteria will be reassessed and the definitive inclusion of the patients will be performed.
  Patients after surgery will go to the anesthetic recovery room and then be admitted to hospital beds, to be discharged within approximately 12 hours.
  1 phone review call will be made per month +/- 30 days in order to assess the safety and satisfaction of the procedure.
  Interventions: Procedure: Hospitalization appendectomy (HA)

INTERVENTIONS:
Procedure: Outpatient (OA) — Patients who are candidates for OA and therefore pre-selected based on the primary data and characteristics of the clinical signs, will be admitted to the surgical observation in charge of our service. The patient will be informed in detail of the intervention to be performed and discharge on an outpatient basis and will sign the informed consent understanding and thus accepting all the information. The patient will undergo surgery using a laparoscopic or open technique with minimal incision.
  Once the appendectomy is performed, all the selection criteria will be reassessed and the definitive inclusion of the patients will be performed. In this case, we will perform the blind randomization of the patients. If all the inclusion requirements for the study are met, and the patient belongs to the OA group (case group), he will be discharged on an outpatient basis from the post-surgical stay unit without requiring hospital admission.
  Arms: Outpatient appendectomy
Procedure: Hospitalization appendectomy (HA) — Patients who are candidates for HA and therefore pre-selected based on the primary data and characteristics of the clinical signs, will be admitted to the surgical observation in charge of our service. The patient will be informed in detail of the intervention to be performed and discharge on an outpatient basis and will sign the informed consent understanding and thus accepting all the information. The patient will undergo surgery using a laparoscopic or open technique with minimal incision.
  Once the appendectomy is performed, all the selection criteria will be reassessed and the definitive inclusion of the patients will be performed. In this case, we will perform the blind randomization of the patients. If all the inclusion requirements for the study are met, and the patient belongs to the case group (HA), he will be admitted in hospital beds.
  Arms: Hospitalization appendectomy

SUMMARY:
This study evaluates the Safety and Efficacy of a outpatient appendectomy. Half of participants will be perform the hospitalization, while the other half will undergo the outpatient appendectomy

DETAILED DESCRIPTION:
Acute appendicitis (AA) is one of the most common causes of acute abdomen and one of the most frequent diagnoses that require urgent surgery worldwide.

Many laparoscopic procedures are currently performed on an outpatient basis.Laparoscopic appendectomy, however, continues to require postoperative hospitalization averaging between 1 and 2 days, at most institutions.

At present ambulatory laparoscopic appendectomy (LA) are gained popularity due to the improved understanding of patient selection criteria, the application of enhanced recovery pathways, and the potential for improving healthcare resource utilization.

There are few studies about to compare the morbidity and readmission rates between ambulatory and conventional LA.

There is a lack of high-quality comparative studies making conclusive recommendations not possible at this time. Based on current data, ambulatory LA may be safe and feasible as compared with conventional LA.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 14 years of age and who provide informed consent to participate in the study.
* Patients with non complicated acute appendicitis requiring and urgent appendectomy (laparoscopic or minimum incision)
* Negative appendicectomy.

Exclusion Criteria:

* Complicated acute appendicitis (abscess, perforated, necrosis and peritonitis)
* Need to place intraoperative drainage.
* Patients with American Society of Anesthesiologists (ASA) >IV.
* Immunosuppressed patients.
* Pregnant.
* Possibility of inflammatory bowel disease.
* No family support.
* No informed consent signature.
* Impossibility to comply with the established follow-up

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 291 (Estimated)
Dates: Start 2019-04-28 (Actual); Primary Completion 2021-04-28 (Estimated); Study Completion 2021-10-28 (Estimated)

PRIMARY OUTCOMES:
Rates of ambulatory appendectomy patients that have ambulatory surgery | 20 months
  Analyze morbidity of appendectomy patients to determine the safety of ambulatory surgery
Rates of readmission of appendectomy patients that had ambulatory surgery | 20 months
  Analyze rates of readmission of appendectomy patients to determine the safety of ambulatory surgery

SECONDARY OUTCOMES:
Prevalence of ambulatory appendectomy patients | 20 months
  Measure the percentage of ambulatory surgery and uncomplicated acute appendicitis vs the percentage of ambulatory surgery in failure patients with the same pathology e.g.
  * Uncontrolled abdominal pain with analgesia.
  * Upper airway discomfort related to intubation that is not controlled with medication.
  * Pain in the back or shoulders in relation to the pneumoperitoneum that are in patients with not controlled with the medication.
  * Hemodynamically abnormal. Uncontrolled bleeding at the level of any of the wounds. Need for reoperation. Need to re-enter or consult the Emergency Service No spontaneous urination.
  * Nausea / vomiting.
  * Oral intolerance.
  * No wandering.
  * Insecurity or fear of the patient at discharge.
Media of time until the total incorporation to the activities of the daily life after appendectomy | 20 months
  To value the time until the total incorporation to the activities of the daily life after appendectomy.
Rates of satisfaction | 20 months
  Measure the degree of satisfaction of our patients with outpatient management after appendectomy, using a satisfaction questionnaire.
Costs of the outpatient regimen versus the hospitalization of patients | 20 months
  Compare the costs of the outpatient regimen versus the hospitalization of patients with uncomplicated acute appendicitis (cost-minimization analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Pareja C Felipe, PhD, Principal Investigator — Hospital Universitario Virgen del Rocio; Padillo R Javier, PhD, Study Director — Hospital Universitario Virgen del Rocio; Durán MC Virginia María, MD, Study Chair — Hospital Universitario Virgen del Rocio
Locations (1):
- Hospital Universitario Virgen Del Rocio, Seville, Spain

REFERENCES:
- [Background] Di Saverio S, Birindelli A, Kelly MD, Catena F, Weber DG, Sartelli M, Sugrue M, De Moya M, Gomes CA, Bhangu A, Agresta F, Moore EE, Soreide K, Griffiths E, De Castro S, Kashuk J, Kluger Y, Leppaniemi A, Ansaloni L, Andersson M, Coccolini F, Coimbra R, Gurusamy KS, Campanile FC, Biffl W, Chiara O, Moore F, Peitzman AB, Fraga GP, Costa D, Maier RV, Rizoli S, Balogh ZJ, Bendinelli C, Cirocchi R, Tonini V, Piccinini A, Tugnoli G, Jovine E, Persiani R, Biondi A, Scalea T, Stahel P, Ivatury R, Velmahos G, Andersson R. WSES Jerusalem guidelines for diagnosis and treatment of acute appendicitis. World J Emerg Surg. 2016 Jul 18;11:34. doi: 10.1186/s13017-016-0090-5. eCollection 2016. PMID 27437029
- [Background] Cash CL, Frazee RC, Abernathy SW, Childs EW, Davis ML, Hendricks JC, Smith RW. A prospective treatment protocol for outpatient laparoscopic appendectomy for acute appendicitis. J Am Coll Surg. 2012 Jul;215(1):101-5; discussion 105-6. doi: 10.1016/j.jamcollsurg.2012.02.024. Epub 2012 May 19. PMID 22609030
- [Background] Aguayo P, Alemayehu H, Desai AA, Fraser JD, St Peter SD. Initial experience with same day discharge after laparoscopic appendectomy for nonperforated appendicitis. J Surg Res. 2014 Jul;190(1):93-7. doi: 10.1016/j.jss.2014.03.012. Epub 2014 Mar 12. PMID 24725679
- [Background] Frazee RC, Abernathy SW, Isbell CL, Isbell T, Regner JL, Smith RD. Outpatient Laparoscopic Appendectomy: Is It Time to End the Discussion? J Am Coll Surg. 2016 Apr;222(4):473-7. doi: 10.1016/j.jamcollsurg.2015.12.053. Epub 2016 Jan 14. PMID 26920990
- [Background] Frazee R, Burlew CC, Regner J, McIntyre R, Peltz E, Cribari C, Dunn J, Butler L, Reckard P, Dissanaike S, Karimi K, Behnfield C, Melo N, Margulies D. Discussion of: "Outpatient laparoscopic appendectomy can be successfully performed for uncomplicated appendicitis: A Southwestern Surgical Congress multicenter trial". Am J Surg. 2017 Dec;214(6):1010-1011. doi: 10.1016/j.amjsurg.2017.10.003. Epub 2017 Oct 5. No abstract available. PMID 29079020
- [Background] Trejo-Avila M, Cardenas-Lailson E, Valenzuela-Salazar C, Herrera-Esquivel J, Moreno-Portillo M. Ambulatory versus conventional laparoscopic appendectomy: a systematic review and meta-analysis. Int J Colorectal Dis. 2019 Aug;34(8):1359-1368. doi: 10.1007/s00384-019-03341-y. Epub 2019 Jul 5. PMID 31273450

DOCUMENTS (1):
  • Informed Consent Form (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT04464382/ICF_000.pdf